CLINICAL TRIAL: NCT00728858
Title: An Open-Label, Randomized Clinical Study to Evaluate the Efficacy, Safety and Genetic Polymorphism of Hypoca(Barnidipine)and Adalat OROS(Nifedipine) in Mild to Moderate Hypertensive Patients
Brief Title: The Efficacy, Safety and Genetic Polymorphism of Hypoca and Adalat OROS in Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 941227
Record Dates: First submitted 2008-05-28; First posted 2008-08-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
Keywords: Hypertension; SNP; Nifedipine; Barnidipine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extract DNA from buffy coat. Test drug concentration in plasma.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Nifedipine and barnidipine act as calcium channel blockers, and are widely prescribed for pressure control of prehypertension and stage 1 hypertension.

CYP3A4 is responsible for the metabolism of nifedipine and nifedipine, while the contribution of CYP3A5 remains ambiguous. This study is aimed to analyze the association between antihypertensive effects of nifedipine as well as barnidipine and single nucleotide polymorphisms of CYP3A4, CYP3A5 and calcium channels.

DETAILED DESCRIPTION:
For each drug, 20 patients will be enrolled. Patients' blood pressure and heart rates will be measured at first visit, followed by visits at week4 , week 8 and week 12. Blood samples will be drawn at week 4 and week 12 for following analyses of drug plasma concentrations. SNPs in CYP3A4, CYP3A5 and calcium channel v 1.2 will be genotyped using SNPstream.

The differences in the decrease of blood pressures and the durg plasma concentrations between genotypes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 20~90 years old patient
* mild to moderate hypertensive patients
* can finish this study
* can sign agreement

Exclusion Criteria:

* severe hypertension
* Heart failure, Arrhythmia
* Liver or kidney failure
* pregnant women
* allergy to dihydropyridines
* attend other clinical trials in past 3 month

Ages: 22 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension patients living in Taiwan
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FU-TIEN CHIANG, Doctor, Study Chair — National Taiwan University Hospital